CLINICAL TRIAL: NCT02111850
Title: A Phase I/II Study of the Treatment of Metastatic Cancer That Expresses MAGE-A3 Using Lymphodepleting Conditioning Followed by Infusion of HLA-DP0401/0402 Restricted Anti-MAGE-A3 TCR-Gene Engineered Lymphocytes and Aldesleukin
Brief Title: T Cell Receptor Immunotherapy Targeting MAGE-A3 for Patients With Metastatic Cancer Who Are HLA-DP0401 Positive
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 140052; 14-C-0052
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Cervical Cancer; Renal Cancer; Urothelial Cancer; Melanoma; Breast Cancer
Keywords: Gene Therapy; Tumor Regression; Immunotherapy; Adoptive Cell Therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Kidney Neoplasms; Melanoma; Breast Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I Experimental Therapy (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + Anti-Melanoma antigen family A, 3 (MAGE-A3)-DP4 T cell receptor (TCR) peripheral blood lymphocytes (PBL) + high-dose aldesleukin
  Interventions: Biological: Anti-MAGE-A3-DP4 T Cell Receptor (TCR) Peripheral Blood Lymphocytes (PBL); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin
- 2/Phase II Experimental Therapy (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + Anti-Melanoma antigen family A, 3 (MAGE-A3)-DP4 T cell receptor (TCR) peripheral blood lymphocytes (PBL) + high-dose aldesleukin
  Interventions: Biological: Anti-MAGE-A3-DP4 T Cell Receptor (TCR) Peripheral Blood Lymphocytes (PBL); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin

INTERVENTIONS:
Biological: Anti-MAGE-A3-DP4 T Cell Receptor (TCR) Peripheral Blood Lymphocytes (PBL) — Day 0: cells will be infused intravenously (i.v.) on the Patient Care Unit over 20 to 30 minutes
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5 % in water (D5W) with Mesna 15 mg/kg /day X 2 days over 1 hour.
  Other Names: Cytoxan
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m^2 /day intravenous piggy-back (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses).
  Other Names: Proleukin

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy for treating patients with metastatic cancer that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying these specific cells with a type of virus (retrovirus) to attack only the tumor cells, and then giving the cells back to the patient. This type of therapy is called gene transfer. In this protocol, we are modifying the patient s white blood cells with a retrovirus that has the gene for anti-Melanoma antigen family A, 3 (MAGE-A3)-DP0401/0402 incorporated in the retrovirus.

Objective:

The purpose of this study is to determine a safe number of these cells to infuse and to see if these particular tumor-fighting cells (anti-MAGE-A3-DP0401/0402 cells) cause tumors to shrink and to be certain the treatment is safe.

Eligibility:

- Adult's age 18-70 with metastatic cancer expressing the MAGE-A3 molecule.

Design:

* Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed
* Leukapheresis: If the patients meet all of the requirements for the study, they will undergo leukapheresis to obtain white blood cells to make the anti-MAGE-A3-DP0401/0402 cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the anti-MAGE-A3-DP0401/0402 cells and aldesleukin. They will stay in the hospital for approximately 4 weeks for the treatment.
* Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking.

DETAILED DESCRIPTION:
Background:

* We have constructed a single retroviral vector that contains both and $ <= chains of a T cell receptor (TCR) that recognizes the DP0401/0402 restricted Melanoma antigen family A, 3 (MAGE-A3) tumor antigen, which can be used to mediate genetic transfer of this TCR with high efficiency.
* In co-cultures with HLA-DP0401/0402 and MAGE-A3 double positive tumors, the anti- MAGE-A3- DP0401/0402 restricted (anti-MAGE-A3-DP4) TCR transduced T cells secreted significant amounts of Interferon gamma (IFN-y) with high specificity.

Objectives:

Primary objectives:

* Determine a safe dose of the administration of autologous cluster of differentiation 4 (CD4) cells transduced with an anti-MAGE-A3-DP0401/0402 restricted (MAGE-A3-DP4) TCR and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen.
* Determine if this approach will result in objective tumor regression in patients with metastatic cancer expressing MAGE-A3-DP4.
* Determine the toxicity profile of this treatment regimen.

Eligibility:

Patients who are human leukocyte antigens (HLA)-DP0401/0402 positive and 18 years of age or older must have

* Metastatic cancer whose tumors express the MAGE-A3-DP4 antigen.
* Previously received and have been a non-responder to or recurred following at least one first line treatment for metastatic disease.

Patients may not have:

- Contraindications for high dose aldesleukin administration.

Design:

* PBMC obtained by leukapheresis will be enriched for CD4 cells and transduced with the retroviral vector supernatant encoding the anti-MAGE-A3-DP4 TCR.
* The study will begin in a standard phase 1 dose escalation. After the maximum tolerated dose (MTD) cell dose has been determined, patients will be enrolled into the phase 2 portion of the trial at the MTD established during the phase 1 portion of the study. In the phase 2 portion, patients will be entered into two cohorts: cohort 1 will include patients with metastatic melanoma; cohort 2 will include patients with renal cancer and other types of metastatic cancer.
* Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumor reactive, TCR gene-transduced peripheral blood mononuclear cells (PBMC) plus intravenous (IV) aldesleukin.
* Patients will undergo complete evaluation of tumor response every 1-6 months until off study criteria are met.
* For each of the 2 strata evaluated in the phase 2 portion, the study will be conducted using a phase 2 optimal design where initially 21 evaluable patients will be enrolled. For each of these two arms of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.
* For both strata, the objective will be to determine if the treatment regimen is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% partial response (PR) + complete response (CR) rate (p1=0.20).

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Metastatic or locally advanced refractory/recurrent cancer that expresses Melanoma antigen family A, 3 (MAGE-A3) as assessed by one of the following methods: Reverse transcription polymerase chain reaction (RT-PCR) on tumor tissue defined as 30,000 copies of MAGE-A3 per 10^6 glyceraldehyde 3-phosphate dehydrogenase (GAPDH) copies, or by immunohistochemistry of resected tissue defined as 10% or greater of tumor cells being 2-3+ for MAGE-A3, or serum antibody reactive with MAGE-A3. Metastatic cancer diagnosis will be confirmed by the Laboratory of Pathology at the National Cancer Institute (NCI).
2. Patients must have previously received prior first line standard therapy (or effective salvage chemotherapy regimens) for their disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred.
3. Patients must be human leucocyte antigen (HLA)-DP4 positive.
4. Patients with 3 or fewer brain metastases that are less than 1 centimeter (cm) in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
5. Greater than or equal to 18 years of age and less than or equal to age 70.
6. Ability of subject to understand and the willingness to sign the Informed Consent Document.
7. Willing to sign a durable power of attorney
8. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1
9. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
10. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be hepatitis C hepatitis C virus (HCV) ribonucleic acid (RNA) negative.
11. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
12. Hematology

    * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim
    * White blood cell (WBC) greater than or equal to 3000/mm^3
    * Platelets count greater than or equal to 100,000/mm^3
    * Hemoglobin > 8.0 g/dl
13. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 2.5 times the upper limit of normal
    * Serum creatinine less than or equal to 1.6 mg/dl
    * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
14. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients must have

    progressing disease after prior treatment. Note: Patients who have previously received ipilimumab and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.
15. Subjects must be co-enrolled in protocol 03-C-0277.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Active systemic infections, (e.g.: requiring anti-infective treatment), coagulation disorders or any other active major medical illnesses
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of any cardiac events including coronary revascularization or ischemic symptoms.
8. Documented left ventricular ejection fraction (LVEF) of less than or equal to 45% testing is required in patients who are

   * greater than or equal to 65 years old
   * Clinically significant atrial and or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or have a history of ischemic heart disease, or chest pain.
9. Documented forced expiratory volume (FEV1) less than or equal to 60% predicted tested in patients with:

   * A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
   * Symptoms of respiratory dysfunction
10. Patients who are receiving any other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-02-07 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgan RA, Dudley ME, Yu YY, Zheng Z, Robbins PF, Theoret MR, Wunderlich JR, Hughes MS, Restifo NP, Rosenberg SA. High efficiency TCR gene transfer into primary human lymphocytes affords avid recognition of melanoma tumor antigen glycoprotein 100 and does not alter the recognition of autologous melanoma antigens. J Immunol. 2003 Sep 15;171(6):3287-95. doi: 10.4049/jimmunol.171.6.3287. PMID 12960359
- [Background] Suri A. Cancer testis antigens--their importance in immunotherapy and in the early detection of cancer. Expert Opin Biol Ther. 2006 Apr;6(4):379-89. doi: 10.1517/14712598.6.4.379. PMID 16548764
- [Background] Robbins PF, Morgan RA, Feldman SA, Yang JC, Sherry RM, Dudley ME, Wunderlich JR, Nahvi AV, Helman LJ, Mackall CL, Kammula US, Hughes MS, Restifo NP, Raffeld M, Lee CC, Levy CL, Li YF, El-Gamil M, Schwarz SL, Laurencot C, Rosenberg SA. Tumor regression in patients with metastatic synovial cell sarcoma and melanoma using genetically engineered lymphocytes reactive with NY-ESO-1. J Clin Oncol. 2011 Mar 1;29(7):917-24. doi: 10.1200/JCO.2010.32.2537. Epub 2011 Jan 31. PMID 21282551
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0052.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2: Arm 1 Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes 1 X 10^7 Cells + Interleukin-2
- Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes 3 X 10^7 Cells + Interleukin-2
- Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes 1 X 10^8 Cells + Interleukin-2
- Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes 3 X 10^8 Cells + Interleukin-2
- Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes 1 X 10^9 Cells + Interleukin-2
- Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes 3 X 10^9 Cells + Interleukin-2
- Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes 1 X 10^10 Cells + Interleukin-2
- Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes 3 X 10^10 Cells + Interleukin-2
- Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes 1 X 10^11 Cells + Interleukin-2
- Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes Maximum Tolerated Dose + Interleukin-2 Other
- Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma: Anti-Melanoma antigen family A, 3-DP4 T Cell Receptor Peripheral Blood Lymphocytes Maximum Tolerated Dose + Interleukin-2 Melanoma
Period: Phase 1 Dose Escalation
Arm/Group | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma
Started | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 6 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant found to be ineligible and not treated. | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 Maximum Tolerated Dose
Arm/Group | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 6 | 5 | 1 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 4 | 5 | 1 | 19
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (0) | 63.2 (0) | 59.3 (0) | 45.9 (0) | 56.9 (1.56) | 27.7 (0) | 44 (0) | 35.2 (0) | 56.03 (8.08) | 41.84 (15.48) | 41.8 (0) | 49.54 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 4 | 1 | 0 | 10
  Male | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 4 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 6 | 4 | 0 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 6 | 5 | 0 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 6 | 5 | 1 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Cell Dose (MTD) of Cluster of Differentiation 4 (CD4) Cells Transduced With an Anti-MAGE-A3-DP0401/0402 Restricted (MAGE-A3-DP4) T Cell Receptor and Aldesleukin
Description: Highest dose at which less than or equal to 1 of 6 patients experienced a dose-limiting toxicity (DLT) (all grade 3 and greater toxicities with the exception of myelosuppression and grade 3 fever, for example) or the highest dose level studied if DLTs are not observed at any of the dose levels.
Time Frame: Before progression to next-higher dose level, at least two weeks
Measure: Number; unit: cells
Groups:
- All Participants on Phase 1: All participants treated on phase 1 dose level 1-9.
Arm/Group | All Participants on Phase 1
Number analyzed (Participants) | 14
cells | 100,000,000,000

2. Primary Outcome: Percentage of Participants Who Have a Clinical Response to Treatment (Objective Tumor Regression)
Description: Percentage of participants who have a clinical response to treatment (objective tumor regression) measured by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.0. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter of target lesions. Progression is at least a 20% increase in the sum of longest diameter of target lesions or the appearance of one or more new lesions. And stable disease is neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: 6 and 12 weeks after cell infusion, then every 3 months x3, then every 6 months x2 years, then per principal investigator discretion, approximately 6 years
Population: One participant was not evaluable because the participant did not receive cell infusion.
Measure: Number; unit: percentage of participants
Arm/Group | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 5 | 1
percentage of participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 100 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22.2 | 20 | 0
  Progression | 100 | 100 | 100 | 100 | 100 | 0 | 100 | 100 | 77.8 | 80 | 100
  Stable Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Adverse Events With Grades ≥1 That Are Possibly, Probably, and/or Definitely Related to Treatment
Description: Aggregate of all adverse events with Grades ≥1 that are possibly, probably, and/or definitely related to treatment. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse events.
Time Frame: 6 weeks after cell infusion
Population: There are no Grade 1 and 5 adverse events related to treatment.
Measure: Number; unit: adverse events
Arm/Group | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 6 | 5 | 1
adverse events
  Grade 2 Anemia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Anorexia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Anxiety - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Blood bilirubin increased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Chills - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Colitis, infectious (e.g., Clostridium difficile) - Probable | 0 | 00 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Cough - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Creatinine increased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Diarrhea - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Dyspnea - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Epistaxis - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Fatigue - Probable | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
  Grade 2 Fever - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 00 | 0 | 2 | 0
  Grade 2 Hemoglobin - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Grade 2 Hypokalemia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Hypophosphatemia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Grade 2 Hypotension - Probable | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
  Grade 2 Hypoxia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Laryngeal hemorrhage - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Leukocytes (total white blood cell) - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Lymphocyte count decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Lymphopenia - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Nasal congestion - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Nausea - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Neutrophils/granulocytes - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Pain: Head/Headache - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Platelet count decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Platelets - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 2 Pruritis - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Psychosis (hallucinations/delusions) - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Purpura - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Rash maculo-papular - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Rash/desquamation - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Rash/desquamation - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Renal/Genitourinary - Other, renal insufficiency - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 2 Wheezing - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 White blood cell decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Grade 3 SGPT (Serum glutamic pyruvic transaminase) - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 SGOT (Serum glutamic oxaloacetic transaminase) - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 SGOT (Serum glutamic oxaloacetic transaminase) - Probable | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Anemia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
  Grade 3 Bilirubin (hyperbilirubinemia) - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Confusion - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Creatinine - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Creatinine - Probable | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Dyspnea (shortness of breath) - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Dyspnea (shortness of breath) - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 3 Febrile neutropenia - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Febrile neutropenia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Febrile neutropenia (fever of unknow origin) - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Febrile neutropenia (fever of unknow origin) - Probable | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1
  Grade 3 Hemoglobin - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 6 | 1
  Grade 3 Hemoglobin - Probable | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Hypophosphatemia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 3 Hypotension - Probable | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 3 Hypoxia - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Hypoxia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Infection - Probable | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 0
  Grade 3 Leukocytes (total white blood cell) - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 3 Lymphocyte count decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
  Grade 3 Lymphopenia - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 3 Neutrophil count decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
  Grade 3 Neutrophils/granulocytes - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Neutrophils/granulocytes - Probable | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 PTT (Partial Thromboplastin Time) - Probable | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Platelet count decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Grade 3 Platelets - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Grade 3 Platelets - Probable | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Potassium, serum-low (hypokalemia) - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Psychosis (hallucinations/delusions) - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Rash/desquamation - Possible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Renal failure - Probable | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Grade 3 Renal/Genitourinary - Other, oliguria - Probable | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Grade 3 Sodium, serum-low (hyponatremia) - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Supraventricular and nodal arrhythmia: Atrial fibrillation - Possible | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Supraventricular and nodal arrhythmia: Atrial fibrillation - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 3 Urine output decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 White blood cell decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
  Grade 4 SGPT (Serum glutamic pyruvic transaminase) - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 SGOT (Serum glutamic oxaloacetic transaminase) - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 Creatinine - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 Dyspnea (shortness of breath) - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 Hemoglobin - Probable | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Hypoxia - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 Leukocytes (total white blood cell) - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 4 Leukocytes (total white blood cell) - Probable | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Lymphocyte count decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Grade 4 Lymphopenia - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 4 | 1
  Grade 4 Lymphopenia - Probable | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 4 Neutrophil count decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 4 Neutrophils/granulocytes - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 3 | 1
  Grade 4 Neutrophils/granulocytes - Probable | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 4 Platelet count decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Grade 4 Platelets - Definite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 2 | 1
  Grade 4 Platelets - Probable | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 4 White blood cell decreased - Probable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

4. Secondary Outcome: Number of Engineered T Cell Receptor (TCR) Cells That Survived at 4 Weeks
Description: T cell receptor (TCR) and vector presence was quantitated in peripheral blood mononuclear cells (PBMC) samples using flow cytometry. It is a process by which cells are suspended in a liquid so they can be counted.
Time Frame: 4 weeks
Population: One participant was not evaluable because the participant did not receive cell infusion.
  One participant was not analyzed because samples was not collected for the Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2" Arm/Group.
Measure: Median (Full Range); unit: cells/uL
Arm/Group | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 6 | 5 | 1
cells/uL | 1.0792 [NA to NA] — There is no full range for a single participant. | 1.9656 [NA to NA] — There is no full range for a single participant. | 2.8676 [NA to NA] — There is no full range for a single participant. |  | 0.17248 [NA to NA] — There is no full range for a single participant. | 2.8 [NA to NA] — There is no full range for a single participant. | 0 [0 to 0] | 6.79 [NA to NA] — There is no full range for a single participant. | 31.9 [2.99 to 142.1] | 84.86 [11.32 to 158.41] | 24.95 [NA to NA] — There is no full range for a single participant.

5. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, an average of 17 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 6 | 5 | 1
Participants | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 6 | 5 | 1

6. Other Pre Specified Outcome: Number of Participants With Dose-limiting Toxicity (DLT)
Description: A dose-limiting toxicity (DLT) is all grade 3 and greater toxicities with the exception of myelosuppression, aldesleukin expected toxicities, expected chemotherapy toxicities, immediate hypersensitivity reactions occurring within 2 hours of cell infusion, grade 3 fever, grade 3 metabolic laboratory abnormalities without significant clinical sequela that resolve within grade 2 within 7 days, and grade 3 autoimmunity that resolves to less than or equal to a grade 2 autoimmune toxicity within 10 days.
Time Frame: Before progression to next-higher dose level, approximately 2 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: All participants treated on phase 1 dose level 1-9.
Arm/Group | Phase 1
Number analyzed (Participants) | 14
Participants | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, an average of 17 months.
Arm/Group | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 0/1 | 1/1 | 1/2 | 0/1 | 1/1 | 1/1 | 5/6 | 4/5 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/2 | 0/1 | 1/1 | 0/1 | 3/6 | 3/5 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 2/2 | 1/1 | 1/1 | 1/1 | 6/6 | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 (N=2) | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 (N=6) | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other (N=5) | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma (N=1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Hemoglobin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Blood
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Urinary tract Not Otherwise Specified (NOS)
Platelets (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (Oliguria) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia: Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Escalation Arm 1, Dose Level 1 - 1 X 10^7 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 2 - 3 X 10^7 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1 Dose Level 3 - 1 X 10^8 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 4 - 3 X 10^8 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 5 - 1 X 10^9 Cells + Interleukin-2 (N=2) | Phase I Dose Escalation Arm 1, Dose Level 6 - 3 X 10^9 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 7 - 1 X 10^10 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 8 - 3 X 10^10 Cells + Interleukin-2 (N=1) | Phase I Dose Escalation Arm 1, Dose Level 9 - 1 X 10^11 Cells + Interleukin-2 (N=6) | Phase 2 Arm 2, Cohort 1- Maximum Tolerated Dose + Interleukin-2 Other (N=5) | Phase 2 Arm 2, Cohort 2 - Maximum Tolerated Dose + Interleukin-2 Melanoma (N=1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hemoglobin (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 3 (8) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Blood
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Lymphocytes count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (11) | 0 (0)
Lymphopenia (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 3 (8) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 3 (5) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PTT (Partial Thromboplastin Time) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain: Head/headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelets count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
Platelets (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 3 (6) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (Oliguria) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (Renal Insufficiency) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia: Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02111850/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT02111850/ICF_001.pdf